CLINICAL TRIAL: NCT03323294
Title: Bioenergetics and Metabolism in Pediatric Populations
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH); University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: BMPP; 206164 (Other: UAMS IRB); 1P20GM109096-01A1 (NIH)
Record Dates: First submitted 2017-09-27; First posted 2017-10-27 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Obesity; Type 2 Diabetes Mellitus; Insulin Resistance
Keywords: Obesity; Pediatric Health; Type 2 Diabetes; Insulin Resistance; Metformin Therapy
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, stool, spit, and cheek cell samples may be retained. The blood sample will be used for bioenergetics and analyte analysis. The sample may be used for future research studies on pediatric nutrition. Urine samples will be collected to measure fat oxidation. The saliva, cheek swab, and stool sample will be used for future research studies on pediatric nutrition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy Lean: Healthy lean individuals (n=20) defined with a Body Mass Index (BMI) ≥ 5th percentile and <85th percentile for age/sex will be recruited. Participants in this cohort will be asked to complete a one-time study visit.
- Healthy Obese: Healthy obese individuals (n=20) defined with a Body Mass Index (BMI) ≥ 95th percentile for age/sex will be recruited. Participants in this cohort will be asked to complete a one-time study visit.
- Obese Insulin Resistant: Obese insulin resistant individuals (n=70) as defined with a Body Mass Index (BMI) ≥ 95th percentile for age/sex and will be recruited. Participants will be asked to complete a total of 2 study visits. The second study visit will occur at 12 months (± 2 weeks) after the initial study visit.
- Type 2 Diabetes or Insulin Resistant: Obese individuals with Type 2 Diabetes or insulin resistance (n=20)

SUMMARY:
The investigators want to learn more about obesity, the development of insulin resistance, and Type 2 Diabetes in children. The investigators will do this through collecting information about children's health and conducting experiments on a variety of samples.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-9 years and Tanner stage as reported by parent no greater than stage 1 OR Age 5 years - 17 years 5 months, diagnosed with type 2 diabetes mellitus or insulin resistance
* Either healthy lean (BMI≥ 5th percentile and <85th percentile for age/sex) or obese (BMI ≥ 95th percentile for age/sex)
* For those with BMI≥ 95th percentile for age/sex, parental verbal confirmation will be obtained that the child had a history of BMI≥ 95th percentile for age/sex for at least six months prior to study enrollment

Exclusion criteria:

* Genetic or physical conditions impacting mobility over past year as determined by the Principal Investigator (PI)
* Having known chronic illnesses/disorders that may independently affect study outcome measures: type 1 diabetes mellitus, neurologic (e.g. epilepsy), developmental (developmental delay, autism spectrum disorder), endocrine (thyroid, Cushing's), hepatic, autoimmune, cardiac and renal disorders. Also, chronic lung disorders except well controlled asthma that does not require permanent use of inhaled/oral steroids
* Taking any of the following medications that can affect study outcome: antipsychotics, thyroid hormone replacement therapy, inhaled/oral steroids, insulin, anabolic drugs (growth hormone replacement therapy and oxandrolone) and stimulants
* BMI<5th percentile for age/sex (classified as underweight based on Centers for Disease Control and Prevention growth charts)
* Subjects determined ineligible by the PI.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Study investigators, research staff, or any qualified personnel will conduct recruitment of study participants using IRB approved advertisement. 175 pre-pubertal children ages 5-9 years old or children diagnosed with type 2 diabetes or insulin resistance ages 5-17 years old will be recruited and may enroll for this study with the goal that 130 subjects stratified across the study groups will complete the study.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Altered circulating blood cell bioenergetics | After completion of all study visits, approximately 2 years.
  The investigators hypothesize that when compared to normal weight or obese insulin sensitive children, obese insulin resistant children will exhibit altered circulating blood cell bioenergetics.
Oxidized plasma redox state | After completion of all study visits, approximately 2 years.
  The investigators hypothesize that when compared to normal weight or obese insulin sensitive children, obese insulin resistant children will exhibit a more oxidized plasma redox state.
Alterations in resting energy expenditure | After completion of all study visits, approximately 2 years.
  The investigators hypothesize that when compared to normal weight or obese insulin sensitive children, obese insulin resistant children will be associated with alterations of decreased resting energy expenditure.
Alterations in fatty acid oxidation | After completion of all study visits, approximately 2 years.
  We hypothesize that when compared to normal weight or obese insulin sensitive children, obese insulin resistant children will be associated with alterations of impaired fatty acid oxidation (FAO).
Poor oxidative capacity | After completion of all study visits, approximately 2 years.
  The investigators hypothesize that poor oxidative capacity over time may distinguish between metabolically healthy obese (MHO) and metabolically unhealthy obese (MUO) phenotypes.
Predicting Type 2 Diabetes development | After completion of all study visits, approximately 2 years.
  The investigators hypothesize that poor oxidative capacity over time may be predictive of Type 2 Diabetes development.
Bioenergetics in Type 2 Diabetes with metformin | 6 months
  The investigators hypothesize that the change in bioenergetics will be improved in obese Type 2 Diabetes children at 6 months of metformin therapy that will be prescribed as part of their clinical care.
Resting Energy Expenditure in Type 2 Diabetes with metformin | 6 months
  The investigators hypothesize that the change in resting energy expenditure will be improved in obese Type 2 Diabetes children at 6 months of metformin therapy that will be prescribed as part of their clinical care.
Fatty Acid Oxidation in Type 2 Diabetes with metformin | 6 months
  The investigators hypothesize that the change in fatty acid oxidation will be improved in obese Type 2 Diabetes children at 6 months of metformin therapy that will be prescribed as part of their clinical care.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Rose, PhD, Study Chair — Arkansas Children's Research Institute; Eugenia Carvalho, PhD, Principal Investigator — Arkansas Children's Nutrition Center
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Yes
The information collected at the study visit, saliva, cheek swabs, blood, urine, and stool samples may be stored indefinitely and may be used for future research studies on pediatric nutrition. Prior to the information collected at the study visit and samples being used for future research studies, the PI will assess the ethics and scientific merit of the proposed research with the samples, and proposed future research will be reviewed by the IRB as may be required. The samples and health information collected for the study visit may be shared with researchers at the University of Arkansas for Medical Sciences, Arkansas Children's Hospital, or Arkansas Children's Research Institute. The samples may be shared with an outside group. The samples will only have a study number and study acronym to maintain confidentiality.
Supporting Information: CSR
Time Frame: The data and samples will be available after all data has been collected for the study and all samples have been processed for the study. Prior to the information collected at the study visit and samples being used for future research studies, the PI will assess the ethics and scientific merit of the proposed research with the samples, and proposed future research will be reviewed by the Institutional Review Board (IRB) as may be required.
Access Criteria: The samples and health information collected for the study visit may be shared with researchers at the University of Arkansas for Medical Sciences, Arkansas Children's Hospital, or Arkansas Children's Research Institute. The samples may be shared with an outside group. The samples will only have a study number and study acronym to maintain confidentiality.

REFERENCES:
- [Background] Mokdad AH, Ford ES, Bowman BA, Nelson DE, Engelgau MM, Vinicor F, Marks JS. Diabetes trends in the U.S.: 1990-1998. Diabetes Care. 2000 Sep;23(9):1278-83. doi: 10.2337/diacare.23.9.1278. PMID 10977060
- [Background] Vincent HK, Innes KE, Vincent KR. Oxidative stress and potential interventions to reduce oxidative stress in overweight and obesity. Diabetes Obes Metab. 2007 Nov;9(6):813-39. doi: 10.1111/j.1463-1326.2007.00692.x. PMID 17924865
- [Background] Civitarese AE, Ravussin E. Mitochondrial energetics and insulin resistance. Endocrinology. 2008 Mar;149(3):950-4. doi: 10.1210/en.2007-1444. Epub 2008 Jan 17. PMID 18202132
- [Background] Hesselink MK, Schrauwen-Hinderling V, Schrauwen P. Skeletal muscle mitochondria as a target to prevent or treat type 2 diabetes mellitus. Nat Rev Endocrinol. 2016 Nov;12(11):633-645. doi: 10.1038/nrendo.2016.104. Epub 2016 Jul 22. PMID 27448057
- [Background] Patti ME, Corvera S. The role of mitochondria in the pathogenesis of type 2 diabetes. Endocr Rev. 2010 Jun;31(3):364-95. doi: 10.1210/er.2009-0027. Epub 2010 Feb 15. PMID 20156986
- [Background] Codoner-Franch P, Pons-Morales S, Boix-Garcia L, Valls-Belles V. Oxidant/antioxidant status in obese children compared to pediatric patients with type 1 diabetes mellitus. Pediatr Diabetes. 2010 Jun;11(4):251-7. doi: 10.1111/j.1399-5448.2009.00565.x. Epub 2009 Sep 16. PMID 19671090
- [Background] Faienza MF, Francavilla R, Goffredo R, Ventura A, Marzano F, Panzarino G, Marinelli G, Cavallo L, Di Bitonto G. Oxidative stress in obesity and metabolic syndrome in children and adolescents. Horm Res Paediatr. 2012;78(3):158-64. doi: 10.1159/000342642. Epub 2012 Oct 10. PMID 23052543
- [Background] Marin MT, Dasari PS, Tryggestad JB, Aston CE, Teague AM, Short KR. Oxidized HDL and LDL in adolescents with type 2 diabetes compared to normal weight and obese peers. J Diabetes Complications. 2015 Jul;29(5):679-85. doi: 10.1016/j.jdiacomp.2015.03.015. Epub 2015 Apr 6. PMID 25881918
- [Background] Matusik P, Prokopowicz Z, Norek B, Olszanecka-Glinianowicz M, Chudek J, Malecka-Tendera E. Oxidative/Antioxidative status in obese and sport trained children: a comparative study. Biomed Res Int. 2015;2015:315747. doi: 10.1155/2015/315747. Epub 2015 Mar 31. PMID 25918709
- [Background] Vehapoglu A, Turkmen S, Goknar N, Ozer OF. Reduced antioxidant capacity and increased subclinical inflammation markers in prepubescent obese children and their relationship with nutritional markers and metabolic parameters. Redox Rep. 2016 Nov;21(6):271-80. doi: 10.1080/13510002.2015.1133035. Epub 2016 Feb 19. PMID 26865084
- [Background] Albuali WH. Evaluation of oxidant-antioxidant status in overweight and morbidly obese Saudi children. World J Clin Pediatr. 2014 Feb 8;3(1):6-13. doi: 10.5409/wjcp.v3.i1.6. eCollection 2014 Feb 8. PMID 25254179
- [Background] Codoner-Franch P, Boix-Garcia L, Simo-Jorda R, Del Castillo-Villaescusa C, Maset-Maldonado J, Valls-Belles V. Is obesity associated with oxidative stress in children? Int J Pediatr Obes. 2010;5(1):56-63. doi: 10.3109/17477160903055945. PMID 19565402
- [Background] Paltoglou G, Fatouros IG, Valsamakis G, Schoina M, Avloniti A, Chatzinikolaou A, Kambas A, Draganidis D, Mantzou A, Papagianni M, Kanaka-Gantenbein C, Chrousos GP, Mastorakos G. Antioxidation improves in puberty in normal weight and obese boys, in positive association with exercise-stimulated growth hormone secretion. Pediatr Res. 2015 Aug;78(2):158-64. doi: 10.1038/pr.2015.85. Epub 2015 May 4. PMID 25938733
- [Background] Santillan LD, Moyano M, Frau M, Flores O, Siewert S, Zirulnick F, Ramirez DC, Gimenez MS. Reduced blood nrf-2 mRNA in local overweight boys at risk of metabolic complications: a study in San Luis City, San Luis, Argentina. Metab Syndr Relat Disord. 2013 Oct;11(5):359-65. doi: 10.1089/met.2012.0155. Epub 2013 Jun 28. PMID 23809001
- [Background] Simoneau JA, Colberg SR, Thaete FL, Kelley DE. Skeletal muscle glycolytic and oxidative enzyme capacities are determinants of insulin sensitivity and muscle composition in obese women. FASEB J. 1995 Feb;9(2):273-8. PMID 7781930
- [Background] Simoneau JA, Bouchard C. Skeletal muscle metabolism and body fat content in men and women. Obes Res. 1995 Jan;3(1):23-9. doi: 10.1002/j.1550-8528.1995.tb00117.x. PMID 7712356
- [Background] Simoneau JA, Kelley DE. Altered glycolytic and oxidative capacities of skeletal muscle contribute to insulin resistance in NIDDM. J Appl Physiol (1985). 1997 Jul;83(1):166-71. doi: 10.1152/jappl.1997.83.1.166. PMID 9216960
- [Background] Simoneau JA, Kelley DE, Neverova M, Warden CH. Overexpression of muscle uncoupling protein 2 content in human obesity associates with reduced skeletal muscle lipid utilization. FASEB J. 1998 Dec;12(15):1739-45. doi: 10.1096/fasebj.12.15.1739. PMID 9837864
- [Background] Kelley DE, Goodpaster B, Wing RR, Simoneau JA. Skeletal muscle fatty acid metabolism in association with insulin resistance, obesity, and weight loss. Am J Physiol. 1999 Dec;277(6):E1130-41. doi: 10.1152/ajpendo.1999.277.6.E1130. PMID 10600804
- [Background] Ritov VB, Menshikova EV, He J, Ferrell RE, Goodpaster BH, Kelley DE. Deficiency of subsarcolemmal mitochondria in obesity and type 2 diabetes. Diabetes. 2005 Jan;54(1):8-14. doi: 10.2337/diabetes.54.1.8. PMID 15616005
- [Background] Ritov VB, Menshikova EV, Azuma K, Wood R, Toledo FG, Goodpaster BH, Ruderman NB, Kelley DE. Deficiency of electron transport chain in human skeletal muscle mitochondria in type 2 diabetes mellitus and obesity. Am J Physiol Endocrinol Metab. 2010 Jan;298(1):E49-58. doi: 10.1152/ajpendo.00317.2009. Epub 2009 Nov 3. PMID 19887598
- [Background] Kelley DE, He J, Menshikova EV, Ritov VB. Dysfunction of mitochondria in human skeletal muscle in type 2 diabetes. Diabetes. 2002 Oct;51(10):2944-50. doi: 10.2337/diabetes.51.10.2944. PMID 12351431
- [Background] Patti ME, Butte AJ, Crunkhorn S, Cusi K, Berria R, Kashyap S, Miyazaki Y, Kohane I, Costello M, Saccone R, Landaker EJ, Goldfine AB, Mun E, DeFronzo R, Finlayson J, Kahn CR, Mandarino LJ. Coordinated reduction of genes of oxidative metabolism in humans with insulin resistance and diabetes: Potential role of PGC1 and NRF1. Proc Natl Acad Sci U S A. 2003 Jul 8;100(14):8466-71. doi: 10.1073/pnas.1032913100. Epub 2003 Jun 27. PMID 12832613
- [Background] Sreekumar R, Halvatsiotis P, Schimke JC, Nair KS. Gene expression profile in skeletal muscle of type 2 diabetes and the effect of insulin treatment. Diabetes. 2002 Jun;51(6):1913-20. doi: 10.2337/diabetes.51.6.1913. PMID 12031981
- [Background] Ten S, Bhangoo A, Ramchandani N, Mueller C, Vogiatzi M, New M, Lesser M, Maclaren N. Resting energy expenditure in insulin resistance falls with decompensation of insulin secretion in obese children. J Pediatr Endocrinol Metab. 2008 Apr;21(4):359-67. doi: 10.1515/JPEM.2008.21.4.359. PMID 18556967
- [Background] De Pergola G, Pannacciulli N, Minenna A, Martina RA, Cannito F, Giorgino R. Fuel metabolism in adult individuals with a wide range of body mass index: effect of a family history of type 2 diabetes. Diabetes Nutr Metab. 2003 Feb;16(1):41-7. PMID 12848304
- [Background] Chacko BK, Kramer PA, Ravi S, Benavides GA, Mitchell T, Dranka BP, Ferrick D, Singal AK, Ballinger SW, Bailey SM, Hardy RW, Zhang J, Zhi D, Darley-Usmar VM. The Bioenergetic Health Index: a new concept in mitochondrial translational research. Clin Sci (Lond). 2014 Sep;127(6):367-73. doi: 10.1042/CS20140101. PMID 24895057
- [Background] Kramer PA, Chacko BK, Ravi S, Johnson MS, Mitchell T, Darley-Usmar VM. Bioenergetics and the oxidative burst: protocols for the isolation and evaluation of human leukocytes and platelets. J Vis Exp. 2014 Mar 27;(85):51301. doi: 10.3791/51301. PMID 24747339
- [Background] Tyrrell DJ, Bharadwaj MS, Van Horn CG, Marsh AP, Nicklas BJ, Molina AJ. Blood-cell bioenergetics are associated with physical function and inflammation in overweight/obese older adults. Exp Gerontol. 2015 Oct;70:84-91. doi: 10.1016/j.exger.2015.07.015. Epub 2015 Jul 29. PMID 26226578
- [Background] Nijhawan S, Richards W, O'Hea MF, Audia JP, Alvarez DF. Bariatric surgery rapidly improves mitochondrial respiration in morbidly obese patients. Surg Endosc. 2013 Dec;27(12):4569-73. doi: 10.1007/s00464-013-3125-y. Epub 2013 Aug 24. PMID 23982645
- [Background] Tyrrell DJ, Bharadwaj MS, Jorgensen MJ, Register TC, Molina AJ. Blood cell respirometry is associated with skeletal and cardiac muscle bioenergetics: Implications for a minimally invasive biomarker of mitochondrial health. Redox Biol. 2016 Dec;10:65-77. doi: 10.1016/j.redox.2016.09.009. Epub 2016 Sep 21. PMID 27693859
- [Background] Bervoets L, Massa G. Classification and clinical characterization of metabolically "healthy" obese children and adolescents. J Pediatr Endocrinol Metab. 2016 May 1;29(5):553-60. doi: 10.1515/jpem-2015-0395. PMID 26910741
- [Background] Munoz-Garach A, Cornejo-Pareja I, Tinahones FJ. Does Metabolically Healthy Obesity Exist? Nutrients. 2016 Jun 1;8(6):320. doi: 10.3390/nu8060320. PMID 27258304
- [Background] Rose S, Frye RE, Slattery J, Wynne R, Tippett M, Melnyk S, James SJ. Oxidative stress induces mitochondrial dysfunction in a subset of autistic lymphoblastoid cell lines. Transl Psychiatry. 2014 Apr 1;4(4):e377. doi: 10.1038/tp.2014.15. PMID 24690598
- [Background] Rose S, Frye RE, Slattery J, Wynne R, Tippett M, Pavliv O, Melnyk S, James SJ. Oxidative stress induces mitochondrial dysfunction in a subset of autism lymphoblastoid cell lines in a well-matched case control cohort. PLoS One. 2014 Jan 8;9(1):e85436. doi: 10.1371/journal.pone.0085436. eCollection 2014. PMID 24416410
- [Result] Santos D, Porter-Gill P, Goode G, Delhey L, Sorensen AE, Rose S, Borsheim E, Dalgaard LT, Carvalho E. Circulating microRNA levels differ in the early stages of insulin resistance in prepubertal children with obesity. Life Sci. 2023 Jan 1;312:121246. doi: 10.1016/j.lfs.2022.121246. Epub 2022 Nov 28. PMID 36455651
- [Result] Barbosa P, Landes RD, Graw S, Byrum SD, Bennuri S, Delhey L, Randolph C, MacLeod S, Reis A, Borsheim E, Rose S, Carvalho E. Effect of excess weight and insulin resistance on DNA methylation in prepubertal children. Sci Rep. 2022 May 19;12(1):8430. doi: 10.1038/s41598-022-12325-y. PMID 35589784
- [Result] Barbosa P, Melnyk S, Bennuri SC, Delhey L, Reis A, Moura GR, Borsheim E, Rose S, Carvalho E. Redox Imbalance and Methylation Disturbances in Early Childhood Obesity. Oxid Med Cell Longev. 2021 Aug 17;2021:2207125. doi: 10.1155/2021/2207125. eCollection 2021. PMID 34457110

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT03323294/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT03323294/ICF_001.pdf